CLINICAL TRIAL: NCT00203528
Title: Divalproex ER vs. Risperidone for Bipolar Disorder With Comorbid Substance Use Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tuscaloosa Research & Education Advancement Corporation (Other)
Collaborators: Abbott (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: TREAC Dual Diagnosis Study; TREAC Dual Diagnosis Study
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2007-03-19 (Estimated); Status verified 2007-03

CONDITIONS: Substance Abuse; Bipolar Depression
Keywords: divalproex sodium; risperidone; dual diagnosis; substance use; bipolar
MeSH Terms: conditions — Substance-Related Disorders; Bipolar Disorder | interventions — Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: divalproex sodium ER
Drug: risperidone

SUMMARY:
The primary objective is to evaluate the safety and efficacy of divalproex extended release (ER) compared to risperidone in the treatment of bipolar disorder with comorbid substance use disorder

DETAILED DESCRIPTION:
Patients will be screened up to seven days at which time the following assessments will be completed: the Structured Clinical Interview for DSM-IV (SCID), general medical history, psychiatric history, physical examination, physicians assessment, and laboratory tests. Patients who are on mood stabilizers and oral neuroleptics prior to study enrollment and are not responding fully to these medications will be tapered off of the medication for a washout period of 48 hours. After the completion of screening, only patients who are determined to be eligible for the study will be randomized to study medication (divalproex or risperidone) in a 1:1 double-blind fashion. Scheduled study visits will occur every two weeks for a total of 12 weeks. Assessments for each visit, from the baseline visit to the week 12 visit are as follows: the Clinical Global Impression (CGI), Global Assessment of Functioning (GAF), Alcohol and Drug Use Inventory, clinician alcohol and drug use scales, self report scales, adverse events, vital signs and weight, concomitant medications, urine drug screen, and study medication accountability. Designated research staff will complete assessments weekly. Investigators will be blinded to laboratory tests completed at week 2, 4, and 12 visits. Patients randomized to Depakote ER will begin 500mg BID on day of randomization and remain on this dose for 5 days, then on day 6 increase to 20mg/kg to achieve valproic acid levels of 80-100 (blinded laboratory reporting). Patients randomized to risperidone, initially start with 2mg QD with an increase to 4mg at day 5 and increase (as tolerated or required) up to 6mg/d.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent for trial participation.
* Male or female patients, ages 19-65.
* Patients must meet DSM-IV criteria for bipolar I or bipolar II disorder (any phase of illness) and concurrent substance use disorder (alcohol or illicit drug abuse or dependence).
* Female patients of childbearing potential must be using a reliable method of contraception. Reliable methods of contraception include hormonal contraceptives (oral contraceptive or long-term injectable or implantable hormonal contraceptive), barrier methods (e.g., condom and diaphragm, condom and foam, condom and sponge), intrauterine devices, and tubal ligation.
* Female patients of child-bearing potential must have a negative urine pregnancy test at screening.
* Patients must not have other serious unstable illnesses and must be otherwise physically stable on the basis of a physical exam, medical history, and the results of blood biochemistry, hematology tests, and a urinalysis.
* Patients must complete at least a 48-hour wash screening/washout period for mood stabilizers and oral neuroleptics.The wash screening/washout period may be completed as an inpatient. If so patient may remain an inpatient as long as necessary. Should the patient become discharged he or she must be able to continue in the study as an outpatient.

Exclusion Criteria:

* Patients with a current DSM-IV diagnosis of schizophrenia or schizoaffective disorder.
* Patients who are legally incompetent
* Receiving any other psychotropic medication within 48 hours of randomization, excluding trazodone for insomnia.
* Patients with Axis I or Axis II diagnosis that in the investigator's opinion, would interfere with compliance or confound interpretation of the results.
* Patients with CNS neoplasm, uncontrolled metabolic, endocrine, demyelinating or progressive neurological disorder, pancreatitis, or urea cycle disorder.
* Patients with a blood chemistries ALT and/or AST value(s) greater than or equal to three times the upper limit of normal prior to randomization.
* Patients with a history of a chronic or acute medical disorder that, in the opinion of the investigator, would confound interpretation of the study results.
* Patients with a medical condition that requires the continuous use of medication that would interfere with the evaluation of safety or efficacy of divalproex ER or risperidone. Patients receiving beta-blockers are excluded unless the dose has been stable for greater than 6 months.
* Patients who have received depot neuroleptic medication within one inter-injection interval of randomization. Patients on depot medications may be included if they are randomized no earlier than the time of their next scheduled depot injection.
* Patients who exhibits signs of drug or alcohol withdrawal at the time of randomization.
* Patients that require the use of naltrexone or disulfiram during the study.
* Patients with a history of previous severe intolerance, idiosyncratic reaction or allergies related to valproate or risperidone.
* Patients with a history of failed treatment on adequate valproate or risperidone therapy for bipolar disorder in the opinion of the investigator.
* Patients who have taken Divalproex DR, Divalproex ER, or risperidone regularly over the 30 days prior to screening/washout. If patients have taken divalproex (either DR or ER) at all in the 30 days prior to screening/washout, a serum valproate level must be done at the time of screening and found to be below the minimum quantifiable limit.
* Women who are pregnant or intends to become pregnant.
* Patient with a platelet count at screening <100,000/mL.
* Patients with serious violent, homicidal, or suicidal ideation.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-01; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
The primary objective is to evaluate the safety and efficacy of divalproex extended release (ER) compared to risperidone in the treatment of bipolar disorder with comorbid substance use disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Lori L Davis, MD, Principal Investigator — Tuscaloosa Veterans Affairs Medical Center
Locations (1):
- Tuscaloosa Research & Education Advancement Corporation, Tuscaloosa, Alabama, United States

REFERENCES:
- [Background] Le Fauve CE, Litten RZ, Randall CL, Moak DH, Salloum IM, Green AI. Pharmacological treatment of alcohol abuse/dependence with psychiatric comorbidity. Alcohol Clin Exp Res. 2004 Feb;28(2):302-12. doi: 10.1097/01.alc.0000113413.37910.d7. PMID 15112938